CLINICAL TRIAL: NCT01940406
Title: The ET and PD Tremor Study - Rainbow Medical Acute Stimulation Evaluation for Tremor Reduction
Brief Title: The Essential Tremor (ET) and Parkinson Disease (PD) Tremor Acute Stimulation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Internal desicions
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-01-001
Record Dates: First submitted 2013-07-16; First posted 2013-09-12 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Essential Tremor; Parkinson Disease
Keywords: Essential Tremor; Parkinson Disease; Electrical Stimulation; Tremor
MeSH Terms: conditions — Essential Tremor; Parkinson Disease; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stimulation procedure (Experimental): Stimulation procedure
  Interventions: Procedure: Stimulation procedure

INTERVENTIONS:
Procedure: Stimulation procedure — Device

SUMMARY:
The current study is designed to test the hypothesis that targeted electrical stimulation will result in upper limb tremor reduction in ET and PD patients.

DETAILED DESCRIPTION:
This study will evaluate the effect of Rainbow Medical's stimulation procedure methodology that will be applied temporarily to patients suffering of tremor.

This will be evaluated by assessment of reduction of tremor using accelerometer measurements, patient tremor evaluation diary, tremor rating scale, and the Unified Parkinson's Disease Rating Scale (UPRDS) part III.In addition,tasks for patient with tremor will be conducted before during and after the treatment. The above measurements will provide data on the stimulation procedure effect as compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Able to Sign written informed consent in Hebrew.
* Patient agrees to attend all treatment procedures and follow-up evaluations and is willing and able to comply with all study requirements.
* Patient with a clinical diagnosis of idiopathic PD, or ET for more than 3 years.
* Significant tremor for at least one upper limb causing distress or disability.
* Patient should be stable on anti-Parkinson's disease or anti-tremor medication for at least one month prior to study enrollment.

Exclusion Criteria:

* Previous participation in another study with any investigational drug or device within the past 90 days.
* Any active implant (cardiac or other).
* Current pregnancy or attempting to get pregnant (female patient).
* Patient has any major illness or medical condition that in the opinion of the physician would interfere with participation in the study.
* Patient with other significant neurological or psychiatric disease other than Parkinson Disease or Essential Tremor.
* Patient has any other condition expect for PD and ET that induce tremor.
* Patient is treated with drug that may induce tremor.
* Patient abuses drugs or alcohol.
* Any previous thalamotomy, pallidotomy or patient who has undergone a DBS procedure.
* Any anticipated need for surgery during the study.
* Any malignancy in the past 2 years.
* Patient has confirmation of diagnosis of a terminal illness associated with survival <12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The severe adverse events rate within the procedure | participants will be followed for the duration of hospital stay, an expected average of 3 weeks

SECONDARY OUTCOMES:
Improvement in tremor symptoms during the procedure | participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Improvement after treatment in ET and PD tremor symptoms in comparison to baseline, as measured by change in:
  * UPDRS part III scale
  * Clinical Tremor Rating Scale
  * Accelerometer values
  * Patient tremor evaluation diary

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Giorini Silfen, PhD, Study Director — BlueWind Medical
Locations (1):
- Department of Neurology, Sheba Medical Center, Tel Litwinsky, Israel